CLINICAL TRIAL: NCT01691014
Title: Formation Of Antibodies And Subsequent Prediction Of Clinical Response In Patients With Rheumatoid Arthritis Treated With Four Tnf Blocking Agents
Status: Terminated | Type: Observational
Why Stopped: The study was terminated on 10DEC2014 due to the inability to enroll the planned number of patients. There were no safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801347
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- adalimumab
  Interventions: Other: non-interventional study
- Etanercept
  Interventions: Other: non-interventional study
- infliximab
  Interventions: Other: non-interventional study
- Certolizumab
  Interventions: Other: non-interventional study

INTERVENTIONS:
Other: non-interventional study — Study with 4 arms/groups with 36 patients per group. In total 144 patients.
  Groups: adalimumab
Other: non-interventional study — Study with 4 arms/groups with 36 patients per group. In total 144 patients.
  Groups: Etanercept
Other: non-interventional study — Study with 4 arms/groups with 36 patients per group. In total 144 patients.
  Groups: infliximab
Other: non-interventional study — Study with 4 arms/groups with 36 patients per group. In total 144 patients.
  Groups: Certolizumab

SUMMARY:
The rationale for this study is to further explore if development of antibodies against TNF-α blocking agents is associated with reduced clinical effect/worsened clinical outcome. An important aspect of the study is to carry out an exploratory analysis of the immunogenicity of the 4 recommended TNF-α blockers in the treatment of RA in Denmark, using the same cell-based assay.

DETAILED DESCRIPTION:
no sampling

ELIGIBILITY:
Inclusion Criteria:

* Subject fulfils criteria for Rheumatoid Arthritis (RA) according to ACR or EULAR criteria.
* Subjects who are planned to start treatment with ADA, ETA, CER or IFX
* Subjects taking a minimum weekly dose of 7.5 mg of methotrexate

Exclusion Criteria:

* Patients with compliance problems
* Patients who have difficulties in reading and understanding local language
* Patients with Juvenile Idiopathic Arthritis (JIA)
* Azathioprine or cyclophosphamide treatment within 6 months before entering into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Rheumatoid Arthritis (RA)
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Denmark (13):
  - Aalborg Universitetshospital Nord/Reumatologisk Afdelning, Aalborg
  - Aarhus Universitetshospital/Reumatologisk Afdelning U, Aarhus C
  - Sydvestjysk Sygehus / Reumatologisk Afdeling, Esbjerg
  - Frederiksberg Hospital / Reumatologisk Afdeling, Frederiksberg
  - Gentofte Hospital, Medicinsk afd. C, Hellerup
  - Hillerod Hospital/Reumatologisk Afdeling, Hillerød
  - Holbaek Sygehus, Holbæk
  - Reumatologisk afd, Kolding
  - Odense Universitets Hospital/Reumatologisk Afdeling C, Odense C
  - Regionshospitalet Randers / Reumatologisk Klinik, Randers NØ
  - Svendborg Sygehus / Medicinsk Afdeling M, Svendborg
  - Vejle Sygehus / Medicinsk Afdeling, Vejle
  - Hospitalsenheden Viborg Reumatologisk Ambulatorium, Viborg

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801347&StudyName=Formation%20of%20Antibodies%20and%20Subsequent%20Prediction%20of%20Clinical%20Response%20in%20Patients%20with%20Rheumatoid%20Arthritis%20Treated%20with%20four%20TNF%20Blockin

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Participants with rheumatoid arthritis (RA) who received adalimumab as per summary of product characteristics (SmPC) during daily clinical practice, were observed prospectively for 12 months.
- Etanercept: Participants with RA who received etanercept as per SmPC during daily clinical practice, were observed prospectively for 12 months.
- Certolizumab: Participants with RA who received certolizumab as per SmPC during daily clinical practice, were observed prospectively for 12 months.
- Infliximab: Participants with RA who received infliximab as per SmPC during daily clinical practice, were observed prospectively for 12 months.
Period: Overall Study
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Started | 8 | 26 | 36 | 9
Completed | 5 | 11 | 25 | 4
Not Completed | 3 | 15 | 11 | 5
Not completed — Premature Termination | 1 | 6 | 0 | 3
Not completed — Other | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 5 | 1 | 1
Not completed — Lack of Efficacy | 2 | 3 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Effectiveness analysis set (EAS) included all participants that provided at least 1 post-baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab | Total
Number analyzed (Participants) | 8 | 26 | 36 | 9 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (6) | 57 (13) | 56 (14) | 51 (11) | 55 (13)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 21 | 23 | 6 | 54
  Male | 4 | 5 | 13 | 3 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-drug Antibodies Formation Levels 6 Months After Initiation of Treatment With Adalimumab, Certolizumab, Etanercept or Infliximab
Description: Anti-drug antibodies to Adalimumab, Certolizumab, Etanercept and Infliximab were to be measured in serum samples using a validated commercially available cell-based reporter-gene assay.
Time Frame: Month 6
Population: Data was not collected since this outcome measure was not analyzed due to premature termination of the study.
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Presence of Active Drugs in Serum 6 Months After Initiation of Treatment With Adalimumab, Certolizumab, Etanercept or Infliximab
Description: Presence of active drugs in serum 6 months after treatment with Adalimumab, Certolizumab, Etanercept and Infliximab were to be measured in serum samples using a validated commercially available cell-based reporter-gene assay.
Time Frame: Month 6
Population: Data was not collected since this outcome measure was not analyzed due to premature termination of the study.
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Correlation Between Formation of Antibodies to Adalimumab, Certolizumab, Etanercept or Infliximab 6 Months After Initiation of Treatment and Disease Activity Score 28 (DAS28) 12 Months After Initiation of Treatment
Description: Association between formation of antibodies to Adalimumab, Certolizumab, Etanercept, Infliximab and DAS28 was to be analyzed using Pearson and Spearman correlations across and within each of the four treatment groups. DAS28-4 was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joint count, C-reactive protein (CRP) in milligram per liter (mg/L) and participant global assessment (PGA) of disease activity (participant rated arthritis activity assessment with total score ranging from 0 [good condition] to 10 [worst condition]; higher score indicates worse condition). DAS28-4 total score range: 0 (no disease activity) to 9.4 (maximum disease activity), higher score indicates more disease activity.
Time Frame: Month 6, 12
Population: Data was not collected since this outcome measure was not analyzed due to premature termination of the study.
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Correlation Between Formation of Antibodies to Adalimumab, Certolizumab, Etanercept or Infliximab 6 Months After Initiation of Treatment and Health Assessment Questionnaire (HAQ) 12 Months After Initiation of Treatment
Description: Association between formation of antibodies to Adalimumab, Certolizumab, Etanercept, Infliximab and HAQ scores was to be analyzed using Pearson and Spearman correlations across and within each of the four treatment groups. HAQ was a self-reported, valid assessment of functional disability in rheumatoid arthritis based on ability of participants to perform daily activities. HAQ total score range: 0 (normal functioning) to 3 (worst functioning), where higher score indicates worse functioning.
Time Frame: Month 6, 12
Population: Data was not collected since this outcome measure was not analyzed due to premature termination of the study.
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Correlation Between Formation of Antibodies to Adalimumab, Certolizumab, Etanercept or Infliximab 6 Months After Initiation of Treatment and Cessation of Therapy Between Month 6 and 12 Visits
Description: Association between formation of antibodies to Adalimumab, Certolizumab, Etanercept and Infliximab and cessation of therapy was to be analyzed. Cessation of therapy between month 6 and month 12 was the time to withdrawal from study due to either adverse events or lack of effect between the 6 month visit and the 12 month visit.
Time Frame: Month 6, 12
Population: Data was not collected since this outcome measure was not analyzed due to premature termination of the study.
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Anti-drug Antibodies Levels 3 and 12 Months After Initiation of Treatment With Adalimumab, Certolizumab, Etanercept or Infliximab
Description: as for outcome 1
Time Frame: Month 3, 12
Population: Data was not collected since this outcome measure was not analyzed due to premature termination of the study.
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Correlation Between the Formation of Anti-drug Antibodies to Adalimumab, Certolizumab, Etanercept or Infliximab and Concomitant Methotrexate Treatment
Description: Association between formation of anti-drug antibodies to Adalimumab, Certolizumab, Etanercept and Infliximab and concomitant Methotrexate treatment (weekly dose of 7.5 milligram) was to be analyzed.
Time Frame: Month 12
Population: Data was not collected since this outcome measure was not analyzed due to premature termination of the study.
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Disease Activity Score Based on 28-Joints Count (DAS28) After Initiation of Treatment With Adalimumab, Certolizumab, Etanercept or Infliximab at Month 3, 6 and 12
Description: DAS28-4 was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joint count, C-reactive protein (CRP) in milligram per liter (mg/L) and participant global assessment (PGA) of disease activity (participant rated arthritis activity assessment with total score ranging from 0 [good condition] to 10 [worst condition]; higher score indicates worse condition). DAS28-4 total score range: 0 (no disease activity) to 9.4 (maximum disease activity), higher score indicates more disease activity. DAS28-4 (CRP) less than or equal to (<=) 3.2 implied low disease activity and greater than (>) 3.2 to 5.1 implied moderate to high disease activity.
Time Frame: Month 3, 6, 12
Population: EAS included all participants that provided at least 1 post-baseline assessment. Here,"n" signifies number of participants evaluable at the specified time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 8 | 26 | 36 | 9
units on a scale
  Month 3 (n= 7, 23, 34, 8) | 3.2 (1.0) | 3.0 (1.1) | 3.0 (1.4) | 3.0 (2.0)
  Month 6 (n= 6, 18, 26, 6) | 2.7 (1.6) | 2.2 (1.1) | 2.4 (1.3) | 1.8 (1.0)
  Month 12 (n= 5, 11, 25, 4) | 2.6 (0.8) | 2.4 (0.8) | 2.5 (1.1) | 2.7 (0.6)
Statistical Analysis 1: Comparison: Adalimumab vs Etanercept vs Certolizumab vs Infliximab; DAS28: Month 3: Continuous variables were compared between treatment groups using one way analysis of variance (ANOVA); Test type: Superiority or Other; p = 0.990, Fisher Exact
Statistical Analysis 2: Comparison: Adalimumab vs Etanercept vs Certolizumab vs Infliximab; DAS28: Month 6: Continuous variables were compared between treatment groups using one way ANOVA; Test type: Superiority or Other; p = 0.586, Fisher Exact
Statistical Analysis 3: Comparison: Adalimumab vs Etanercept vs Certolizumab vs Infliximab; DAS28: Month 12: Continuous variables were compared between treatment groups using one way ANOVA; Test type: Superiority or Other; p = 0.980, Fisher Exact

9. Secondary Outcome: Health Assessment Questionnaire (HAQ) Score After Initiation of Treatment With Adalimumab, Certolizumab, Etanercept or Infliximab at Baseline, Month 3, 6 and 12
Description: HAQ was a self-reported, valid assessment of functional disability in rheumatoid arthritis based on ability of participants to perform daily activities. HAQ total score range: 0 (normal functioning) to 3 (worst functioning), where higher score indicates worse functioning.
Time Frame: Baseline, Month 3, 6, 12
Population: EAS included all participants that provided at least 1 post-baseline assessment. Here, "n" signifies number of participants evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Number analyzed (Participants) | 8 | 26 | 36 | 9
units on a scale
  Baseline (n= 8, 26, 36, 9) | 1.1 (0.6) | 1.2 (0.6) | 1.2 (0.7) | 1.1 (0.5)
  Month 3 (n= 7, 23, 34, 8) | 0.8 (0.6) | 0.9 (0.7) | 0.8 (0.7) | 1.2 (0.8)
  Month 6 (n= 6, 18, 26, 6) | 0.8 (0.2) | 0.6 (0.6) | 0.7 (0.6) | 0.8 (0.7)
  Month 12 (n= 5, 11, 25, 4) | 0.7 (0.4) | 1.0 (0.8) | 0.6 (0.6) | 0.8 (0.7)
Statistical Analysis 1: Comparison: Adalimumab vs Etanercept vs Certolizumab vs Infliximab; HAQ: Baseline: Continuous variables were compared between treatment groups using one way ANOVA; Test type: Superiority or Other; p = 0.945, Fisher Exact
Statistical Analysis 2: Comparison: Adalimumab vs Etanercept vs Certolizumab vs Infliximab; HAQ: Month 3: Continuous variables were compared between treatment groups using one way ANOVA; Test type: Superiority or Other; p = 0.458, Fisher Exact
Statistical Analysis 3: Comparison: Adalimumab vs Etanercept vs Certolizumab vs Infliximab; HAQ: Month 6: Continuous variables were compared between treatment groups using one way ANOVA; Test type: Superiority or Other; p = 0.896, Fisher Exact
Statistical Analysis 4: Comparison: Adalimumab vs Etanercept vs Certolizumab vs Infliximab; HAQ: Month 12: Continuous variables were compared between treatment groups using one way ANOVA; Test type: Superiority or Other; p = 0.390, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline upto 12 months
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participants may have experienced both a serious and non-serious event during the study.
Arm/Group | Adalimumab | Etanercept | Certolizumab | Infliximab
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/26 | 2/36 | 0/9
Other Adverse Events (participants affected / at risk) | 2/8 | 13/26 | 6/36 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=8) | Etanercept (N=26) | Certolizumab (N=36) | Infliximab (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Adenocarcinoma of esophagus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=8) | Etanercept (N=26) | Certolizumab (N=36) | Infliximab (N=9)
Thrombopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Periumbilical pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Feeling unwell (General disorders) | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0
Therapeutic product ineffective (General disorders) | 0 | 1 | 0 | 0
Polyp (General disorders) | 0 | 0 | 0 | 1
Foreign body reaction (General disorders) | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Allergy NOS (Immune system disorders) | 0 | 0 | 0 | 1
Cold (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Infection localised (Infections and infestations) | 1 | 0 | 0 | 0
Nose infection NOS (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Cold sores lip (Infections and infestations) | 0 | 1 | 0 | 0
Flu symptoms (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Elevated liver enzymes (Investigations) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema aggravated (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension arterial (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis leg (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to premature termination of the study, the primary objective and few of the secondary objectives for the study were not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.